CLINICAL TRIAL: NCT07347561
Title: Myoelectric and Bionic Hands in Upper Limb Amputations: A Comparison of Body Image, Function and User Satisfaction
Brief Title: A Comparison of Myoelectric and Bionic Hands
Status: Recruiting | Type: Observational
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Güllü Aydın Yağcıoğlu, Asst. Prof, Gulhane School of Medicine
Other Study IDs: O&P
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-11

CONDITIONS: Amputation; Upper Limb Amputation; Prosthesis
Keywords: Amputation; bionic hand; myoelectric hand; prosthesis; trans-humeral; trnas-radial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bionic Prosthetic Hand Group: Participants use advanced myoelectric prosthetic hands with multi-articulating structures and enhanced control features designed to improve functional performance.These devices are designed to enhance hand function, dexterity, and user interaction beyond conventional myoelectric control.
- Myoelectric Prosthetic Hand Group: Participants in this group are individuals with upper limb amputation who use a myoelectric prosthetic hand controlled by surface electromyographic signals from residual limb muscles. These devices provide electrically powered hand movement and basic grasp functions without advanced bionic or sensor-integrated features.

SUMMARY:
This observational study aims to compare myoelectric and bionic hands in terms of upper extremity function, body image and satisfaction.

The main questions it aims to answer are:

- Does upper extremity function differ between bionic and myoelectric hands?

The main questions it aims to answer are:

Does upper extremity function differ between bionic and myoelectric hands?

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years
* Individuals with unilateral upper limb amputation
* Regular use of a prosthetic device for at least 6 months
* Use of a semi-electronic elbow joint prosthetic component
* Ability to understand and complete study assessments

Exclusion Criteria:

* Presence of bilateral or multiple limb amputations
* Proximal upper limb amputation at the shoulder level or above
* Coexisting neurological or orthopedic disorders that may affect upper limb function or study outcomes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included individuals aged 8-65 who had undergone upper limb amputation.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Upper Limb Functionol Index-15 | Baseline
  The Upper Limb Functional Index-15 (ULFI-15) is a 15-item patient-reported outcome measure used to assess functional limitations related to the upper extremity. It evaluates difficulties in daily activities, movement, and functional performance of the upper limb. Higher scores indicate greater functional limitation.
Amputee Body Image Scale | Baseline
  The Amputee Body Image Scale (ABIS) is a self-reported questionnaire designed to assess body image perception and body-related concerns in individuals with limb amputation. It measures the psychological impact of amputation on body image, with higher scores reflecting greater body image disturbance.
Orthotics and Prosthetics Users' Survey | Baseline
  The Orthotics and Prosthetics Users' Survey (OPUS) is a validated patient-reported outcome measure used to evaluate functional status, satisfaction, and quality of life in individuals using orthotic or prosthetic devices. It assesses the user's perceived functional ability and satisfaction with their prosthetic device and related services.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Gülhane Faculty of Health Sciences, Ankara, Keçiören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carey SL, Lura DJ, Highsmith MJ; CP; FAAOP. Differences in myoelectric and body-powered upper-limb prostheses: Systematic literature review. J Rehabil Res Dev. 2015;52(3):247-62. doi: 10.1682/JRRD.2014.08.0192. PMID 26230500
- [Result] Kannenberg, A., Lundstrom, R., Hibler, K. D., & Johnson, S. S. (2023). Differences in two multiarticulating myoelectric hands for facilitating activities of daily living in individuals with transradial amputation: a cross-sectional study. JPO: Journal of Prosthetics and Orthotics, 35(1), 38-43.